CLINICAL TRIAL: NCT06895304
Title: Effects of Inspiratory Muscle Fatigue and Warm-up on Respiratory Variables, Handgrip Strength, and Walking Capacity in Sedentary Older Adults: A Randomized Clinical Trial.
Brief Title: Effects of Inspiratory Muscle Fatigue and Warm-up on Respiratory Variables, Handgrip Strength, and Walking Capacity in Sedentary Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 018
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Sedentary; Healthy
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: the outcome assessor will not know in which group is each participant, and the investigator will receive the data without knowing which data is from which group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inspiratory muscle fatigue group (Experimental): The EG (fatigue group) will perform the diaphragmatic fatigue protocol using a specific inspiratory endurance test, in which volunteers, one-on-one, and in a single session, will breathe against submaximal inspiratory loads equivalent to 60% of their MIP (Maximum Inspiratory Pressure) through a threshold valve device. The participants will follow a free pattern of breathing until they are unable to establish flow during at least 3 maximum inspiratory efforts.
  Interventions: Device: inspiratory muscle training
- Control group (No Intervention): they will not receive any intervention. Just sit and wait the same amount of time that the intervention and the activation group needs to finish their protocol (around 10 minutes)
- Inspiratory muscle activation group (Active Comparator): The activation group will perform the protocol of 2 sets of 30 repetitions at 15% of their MIP, one-on-one, and in a single session, breathing against submaximal inspiratory loads using a threshold valve device. The participants will follow a free pattern of breathing until complete the protocol.
  Interventions: Device: inspiratory muscle training

INTERVENTIONS:
Device: inspiratory muscle training — The subjects will perform deep inspirations against a threshold device with varying resistances to observe the effect on the diaphragm and the musculature of the upper limbs.
  Other Names: Inspiratory muscle fatigue
  Arms: Inspiratory muscle fatigue group
Device: inspiratory muscle training — The subjects will perform deep inspirations against a threshold device with varying resistances to observe the effect on the diaphragm and the musculature of the upper limbs.
  Other Names: Inspiratory muscle activation
  Arms: Inspiratory muscle activation group

SUMMARY:
Respiratory muscle training represents an effective method increasingly utilized in both sports and healthcare domains, employing various devices, among which threshold devices are prominent. The aim of this study is to determine the relationship between inspiratory muscle fatigue or warm-up and muscular strength in upper and lower limbs, in sedentary older adults, as well as the association between such fatigue and other variables, including maximal inspiratory pressure, diaphragmatic ultrasonography, functionality and handgrip strength.

According to our hypothesis, the execution of a protocol inducing inspiratory muscle fatigue or activation in sedentary older adults could influence muscular strength, respiratory function and exercise capacity.

In this study, subjects will be divided into three groups: the fatigue group , the activation group and the control group.

Measurements of variables, such as maximal inspiratory pressure, diaphragmatic strength (ultrasound image) and functional capacity, will be conducted.

DETAILED DESCRIPTION:
This is a randomized control trial. The fatigue group (EG) will perform the inspiratory muscle fatigue protocol using a specific inspiratory endurance test, in which volunteers, one-on-one, and in a single session, will breathe against submaximal inspiratory loads equivalent to 60% of their Maximum Inspiratory Pressure (MIP) through a threshold valve device. The participants will follow a free pattern of breathing until they are unable to establish flow during at least 3 maximum inspiratory efforts.

The activation group (AG) will perform the protocol of 2 sets of 30 repetitions at 15% of their MIP, one-on-one, and in a single session, using a threshold valve device.

The control group will do a seat and wait.

The interventions will be supervised by a physiotherapist. The primary outcomes will be

Walking capacity will be assessed using the 6 minutes walking test (6MWT) immediately before intervention and immediately after intervention Respiratory muscle strength will be assessed using a respiratory pressure meter or manometer designed, and with ultrasound image measuring the cross sectional area of the diaphragm at 8-9th rib level and speed of contraction with a deep and fast inspiratory manoeuver. This will be done immediately before intervention and immediately after intervention Handgrip strength will be assessed using a handgrip dynamometer. This will be done immediately before intervention and immediately after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being over 60 years old.
* Physical independence in terms of gait and transfers
* Engaging in less than 150 minutes of physical activity per week.

Exclusion Criteria:

* Having any pathology that prevents the performance of physical activity.
* Subjects with impaired cognitive abilities.
* Subjects with tympanic perforation or middle-inner ear pathology.
* Subjects with chronic respiratory, cardiac, renal, or metabolic pathology..
* Subjects who have undergone lower limb surgery within the past 12 months.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | Immediately before intervention and immediately after intervention
  It will be assessed using a MicroRPM® (MicroMedical, UK).
  Maximum Inspiratory Pressure (MIP): The person will be instructed to take a maximal deep breath in, and then exhale to residual volume. After that, they will be asked to inhale forcefully against the resistance provided by the MicroRPM®. This measures the strength of the inspiratory muscles.
  The measures will be expressed in cmH2O.
Diaphragmatic thickness and thickening fraction | Immediately before intervention and immediately after intervention
  Diaphragmatic thickness and thickening fraction The linear array probe with a frequency of 3.0-10 megahertz (MHz) is placed perpendicularly to chest wall close to the mid-axillary line which is between the 8th and 10th intercostal space. The thickness of diaphragm is measured at the end of expiration and maximum inspiration for three times and the average values were recorded.
  The measures will be expressed in centimeters.
Diaphragm movement curve | Immediately before intervention and immediately after intervention
  The convex array probe with a frequency of 1.5-4.6 MHz is placed below the midclavicular line of the right costal margin in longitudinal scanning plane. The liver was used as an inspection window, and the probe was pointed toward the cephalic side. The ultrasound bundle is perpendicular to the posterior third of the right diaphragm. M-mode ultrasound is used to record the diaphragmatic movement curve during quiet breathing (QB) and deep breathing (DB).
  The measures will be expressed in milliseconds.

SECONDARY OUTCOMES:
6 minutes walking test | Immediately before intervention and immediately after intervention
  The 6-Minute Walk Test (6MWT) is a functional cardiorespiratory assessment that measures the maximum distance a subject can walk in six minutes. The patient will be instructed to walk at the fastest possible pace along a 30-meter corridor. The therapist will accompany the patient throughout the test, and the use of assistive devices and/or external oxygen supplementation will be permitted if necessary.
  The measures will be expressed in meters.
Handgrip strength | Immediately before intervention and immediately after intervention
  The recommendations of the American Society of Hand Therapists will be followed: the subject will be positioned with the shoulder in adduction and neutral rotation, the elbow flexed at 90°, the forearm in a neutral position, and the wrist positioned between 0° and 30° of extension.
  Three maximum grip strength measurements will be performed on the dominant hand, with one-minute rest intervals between trials, selecting the highest value.
  Handgrip strength dynamometry will be conducted using a JAMAR dynamometer (Lafayette Instrument, Lafayette, IN, USA).
  The measures will be expressed in kilograms

IPD SHARING:
Plan to Share IPD: Undecided